CLINICAL TRIAL: NCT05648747
Title: Factors Associated With an Unfavorable Clinical Course in Hospitalized Patients With Pelvic Inflammatory Disease in Post Covid 19 Era: a Multicentric Retrospective Cohort Study
Brief Title: Pelvic Inflammatory Disease in COVID-19 Era
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Università degli Studi di Ferrara (Other)
Responsible Party: Principal Investigator, Gennaro Scutiero, MD, Università degli Studi di Ferrara
Other Study IDs: 826/2022/Oss/AOUFe
Record Dates: First submitted 2022-12-09; First posted 2022-12-13 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-12

CONDITIONS: Pelvic Inflammatory Disease
MeSH Terms: conditions — Pelvic Inflammatory Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Complicated Pelvic Inflammatory Disease: The development of complicated Pelvic Inflammatory Disease diagnosed during laparoscopy or by pre-operative image study
  Interventions: Other: impact of COVID-19 on Health-Seeking Behaviors
- Non-Complicated Pelvic Inflammatory Disease: No development of complicated Pelvic Inflammatory Disease diagnosed during laparoscopy or by pre-operative image study
  Interventions: Other: impact of COVID-19 on Health-Seeking Behaviors

INTERVENTIONS:
Other: impact of COVID-19 on Health-Seeking Behaviors — The impact of the coronavirus disease 2019 (COVID-19) pandemic on medical services is overwhelming due to limited medical resources. During its initial surge in 2020, Italy's government rapidly established diverse public actions, which helped maintain the medical supply. However, whether the fear of being infected with COVID-19 interfered with health-seeking behavior (HSB) remains unclear. Therefore, this study aimed to elucidate whether pelvic inflammatory disease rates were affected by the COVID-19 pandemic.

SUMMARY:
The goal of this retrospective cohort study is to to scrutinize the impact of coronavirus disease 2019 (COVID-19) on incidence, demography and patient characteristics in Pelvic Inflammatory Disease comparing with the equal time duration, before and after lockdown was initiated in the country.

The main aim of this study was to compare the demographic and clinical parameters between two cohorts before the onset of lockdown and within the pandemic.

ELIGIBILITY:
Inclusion Criteria:

Pelvic Inflammatory disease

Exclusion Criteria:

Pregnancy Oncologic disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A retrospective analysis of pelvic inflammatory disease in women was performed between March 8, 2020 and March 31, 2022 (COVID-19 period). The control period was collected between January , 2020 and December 31, 2019.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-01-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of pelvic inflammatory disease (PID) | baseline, pre-surgery
  The primary outcome measure was the occurrence of PID defined as abscess observed in computed tomography or a description of gangrenous salpingitis assessed by pathological reports.

CONTACTS AND LOCATIONS:
Locations (1):
- Section of Obstetrics and Gynecology, Department of Morphology, Surgery and Experimental Medicine, University of Ferrara, Ferrara, Italy, Ferrara, Italy

IPD SHARING:
Plan to Share IPD: No